CLINICAL TRIAL: NCT05321576
Title: Comparison of ESPB With Opioid-free Anesthesia and Standardopioid Anesthesia in Patients Who Underwent Lobectomy With VATS Method: a Randomized Controlled Study.
Brief Title: Opioid-free Anesthesia With ESPB in VATS Operation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Meliha Orhon, assistant professor, Marmara University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 09.2022.100
Record Dates: First submitted 2022-03-03; First posted 2022-04-11 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-03

CONDITIONS: Opioid Use
MeSH Terms: interventions — Methods

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- erector spinae plane block group (Active Comparator): Before this process, it will be produced from the bupivacaine plan, which will be made by entering unilaterally 3 cm lateral in the ultrasound to be made from a work section that will be made before the shipment and by lidocaine.
  Interventions: Procedure: Erector spinae plane block (ESPB) technique without opioid use
- control group (Active Comparator): give opiod in this group of patients
  Interventions: Procedure: Erector spinae plane block (ESPB) technique without opioid use

INTERVENTIONS:
Procedure: Erector spinae plane block (ESPB) technique without opioid use — Local anesthetic injection to the erector spinae muscle plane at T5 level on the operation side.
  Other Names: Standard opioid anesthesia

SUMMARY:
Patients with an ASA score of 3 and below, who will undergo lobectomy with video-assisted thoracic surgery (VATS) method, and who gave informed consent will be included in this study. Patients with contraindications for the application of either of the two methods, with known chronic pain, opioid use, local anesthetic allergy, spinal deformity or mental or psychiatric problems that prevent cooperation, those taking anticoagulants, and those with infection at the injection site will not be included in the study. In addition, patients in the ESPB group who required intraoperative opioids, patients who failed ESPB, and patients who underwent open surgery in both groups will not be included in the analysis. Patients who agree to participate in the study will be randomly assigned to one of the study's opioid-free anesthesia and ESPB (erector spina plan block) (Group 1) or standard opioid (Group 2, control) anesthesia groups. Randomization will be at the ratio of 1:1 and will be done by the closed envelope method. Beforehand, a piece of paper with the name of one of the two groups will be placed inside the envelopes and the envelopes will be closed and mixed. A closed envelope will be drawn at random before the procedure for each patient, and procedures will be carried out according to the group specified on the paper.

DETAILED DESCRIPTION:
Group 1 (opioid-free ESPB) Before induction of anesthesia, patients in this group will undergo ultrasound guidance in a sitting position on the operating table, and an erector spina plan block will be performed with bupivacaine and lidocaine, by entering unilaterally (to the side to be operated) 3 cm lateral to the T5 spinous process. Under standard monitoring (ECG, non-invasive blood pressure, and finger oxygen saturation), anesthesia induction will be performed with propofol (2 mg/kg), ketamine 2 mg/kg, and rocuronium 0.6 mg/kg. Bispectral index (BIS) and analgesia nociception index (ANI) monitoring will be started immediately after intubation. Patients will not take any opioids throughout the surgery and will be infused with dexmedetomidine instead. Dexmedetomidine infusion will be started at a dose of 0.4 microgram/kg/hour, BIS < 50 and the dose of dexmedetomidine will be adjusted so that ANI > 50. Patients for whom dexmedetomidine could not be sufficiently effective and opioid use became mandatory will not be included in the analysis. Before postoperative awakening, patients were given 1 g i.v. paracetamol will be given.

Group 2 (standard anesthesia with opioid) Under standard monitoring (ECG, non-invasive blood pressure, and finger oxygen saturation), anesthesia induction will be performed with propofol (2 mg/kg), remifentanil 1 microgram/kg, and rocuronium 0.6 mg/kg. Bispectral index (BIS) and analgesia nociception index (ANI) monitoring will be started immediately after intubation. Patients will receive an infusion of remifentanil throughout the surgery. Remifentanil infusion will be started at a dose of 0.5 microgram/kg/hour, and the dose of remifentanil will be adjusted so that BIS < 50 and ANI > 50. Before postoperative awakening, patients were given 1 g i.v. paracetamol will be given.

Perioperative clinical and demographic data of each patient will be collected: age, gender, diagnosis, operation, ASA status, duration of surgery, duration of anesthesia. Intraoperatively, heart rate, blood pressure, ANI and BIS measurements will be made and recorded in all patients at 15-minute intervals. In addition, the total intraoperative opioid dose (Group 2) and dexmedetomidine (Group 1) dose will be recorded.

Post-awakening pain will be assessed and recorded using a visual analog scale (VAS), then patient-controlled analgesia (PCA) will be initiated, with all patients locked in 15 minutes and given 4 mg of morphine at each application by the patient. Pain assessment will be done with VAS at 6, 12, 24 and 48 hours postoperatively. In the postoperative period, the amount of morphine administered by PCA (in the first and second 24 hours) and the required additional analgesics (tramadol, paracetamol, etc.) will be recorded. Groups will be compared for primary outcome measure and secondary outcome measure.

Although neuropathic pain after VATS is less than the thoracotomy approach, it can still pose a significant postoperative problem. Pain management after VATS is especially important to prevent respiratory complications. However, intraoperative or postoperative excess morphine consumption will also negatively affect postoperative recovery after thoracic surgery. It has been shown that opioid-free anesthesia can reduce the need for morphine and reduce related complications.

In the ultrasound-guided erector spina plan block technique, which is a regional anesthesia technique that has been defined recently, local anesthetic is injected into the erector spina muscle and facial plane and spreads in the caudal and cranial directions. This technique has been successfully used as a postoperative analgesia or intraoperative regional anesthesia technique in areas such as thoracic surgery and trauma, breast surgery, abdominal surgery, and extremity surgery. Erector spina plane block or other block methods have been mostly used for postoperative analgesia after VATS, and they have been shown to provide effective postoperative analgesia and reduce morphine consumption. However, data on the use of ESPB or other block techniques for anesthesia during VATS are limited. Opioid-free anesthesia with the help of ESPB may help recovery by reducing total and postoperative morphine consumption.

The aim of this study is to compare opioid-free anesthesia with ultrasound-guided ESPB in patients who underwent lobectomy with VATS, with standard opioid-containing anesthesia in terms of postoperative morphine requirement, as well as intraoperative variables, postoperative pain management and postoperative recovery, and complications.

ELIGIBILITY:
Inclusion Criteria:

* lobectomy with video-assisted thoracic surgery (VATS) method
* ASA score of 3 and below
* willing to be included

Exclusion Criteria:

* chronic pain
* current opioid use
* local anesthetic allergy
* spinal deformity or mental or psychiatric problems that prevent cooperation
* anticoagulant use
* infection at the injection site

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2022-04-10 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Opioid consumption | the first 48 hours after surgery
  measurement of postoperatif opioid requirement and consumption

CONTACTS AND LOCATIONS:
Overall Officials: MELIHA ORHON ERGUN, Principal Investigator — Marmara University
Locations (1):
- Marmara University, Istanbul, Maltepe, Turkey (Türkiye)